CLINICAL TRIAL: NCT02841657
Title: 3D vs 2D Colorectal Resections and Valuation of Visual Load of Surgeons
Brief Title: 3D Laparoscopy Versus 2D Laparoscopy
Acronym: Lap3D
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Casa di Cura Dott. Pederzoli (Other)
Responsible Party: Principal Investigator, Marco Inama, General Surgeon, Casa di Cura Dott. Pederzoli
Other Study IDs: 3Dvs2D
Record Dates: First submitted 2016-07-18; First posted 2016-07-22 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Cancer; Inflammatory Bowel Disease
Keywords: 3 Dimensional Laparoscopy; Visual work load; Nasa Task Load Index; Simulator Sickness Questionnaire
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
* To compare surgical and oncological outcomes in patients underwent to colorectal resection with 3D vs 2D laparoscopic technique.
* To evaluate the visual overload in surgeons using 3D laparoscopic technique.

DETAILED DESCRIPTION:
3 Dimensional (3D) Camera system is a new technique introduced into laparoscopic surgery field, adding the depth perception. Even if in the first 2000' the old 3D camera had negative results in terms of quality of images, thanks to technological progress the new 3D systems have reached high quality.

This new technology has been widely tested in pelvic trainer, not yet in live surgery. Moreover effects on surgeons visual work load are unknown.

Aim of the present study is to evaluate the potential superiority of 3D laparoscopic technique on 2D one in terms on postoperative complications and oncological radicality (in case of neoplastic disease).

Secondary aim is to study the possible major visual stress on surgeons brain caused by 3D camera rather than 2D videos.

ENROLLMENT All patients affected by neoplastic or inflammatory colorectal disease are enrolled in the study.

Preoperative, intraoperative e postoperative data are collected dividing all the patients according the camera system used during the operation: 2D group vs 3D group.

Preoperative data: sex, age, date of birth, id, date of admission, past medical history Intraoperative data: date of surgery, pathology, site of pathology, type of surgery and duration, intraoperative blood loss, other intraoperative problems, loop ileostomy, colostomy, drain positioning, intensive care unit admission Postoperative data (at 30th postoperative day): complications according to Dindo-Clavien scale (Dindo-Clavien classification of surgical complications), type of complications, transfusion, reoperation, other treatments, histology specimen report.

At the end of every operation, the 1st surgeon has to fill in the NASA (The National Aeronautics and Space Administration) task load index and the Simulator Sickness questionnaire.

Number of participants: 350 Years necessary: 2

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer with or without preoperative radio e chemiotherapy
* inflammatory bowel disease affected colon and rectum that need surgery

Exclusion Criteria:

* patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients affected by neoplastic and inflammatory disease of colorectal tract can be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | through study completion, an average of 2 years
  The postoperative course is evaluate in all patients undergone to colorectal laparoscopic surgery and classified according to the Dindo-Clavien scale at 30 days after surgery (Dindo-Clavien classification of surgical classification).

SECONDARY OUTCOMES:
Oncological radicality | through study completion, an average of 2 years
  The R0/R1 rate is evaluate in patients undergone to 3 dimensional or 2 dimensional laparoscopic colorectal surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Inama, MD PhDs, Principal Investigator — Hospital "Dott. Pederzoli"
Locations (1):
- Hospital "Dott. Pederzoli", Peschiera del Garda, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Poudel S, Kurashima Y, Watanabe Y, Ebihara Y, Tamoto E, Murakami S, Nakamura T, Tsuchikawa T, Okamura K, Shichinohe T, Hirano S. Impact of 3D in the training of basic laparoscopic skills and its transferability to 2D environment: a prospective randomized controlled trial. Surg Endosc. 2017 Mar;31(3):1111-1118. doi: 10.1007/s00464-016-5074-8. Epub 2016 Jun 28. PMID 27351662
- [Result] Sinha RY, Raje SR, Rao GA. Three-dimensional laparoscopy: Principles and practice. J Minim Access Surg. 2017 Jul-Sep;13(3):165-169. doi: 10.4103/0972-9941.181761. PMID 27143695
- [Result] Shakir F, Jan H, Kent A. 3D straight-stick laparoscopy versus 3D robotics for task performance in novice surgeons: a randomised crossover trial. Surg Endosc. 2016 Dec;30(12):5380-5387. doi: 10.1007/s00464-016-4893-y. Epub 2016 Apr 8. PMID 27059971
- [Result] Sakata S, Watson MO, Grove PM, Stevenson AR. The Conflicting Evidence of Three-dimensional Displays in Laparoscopy: A Review of Systems Old and New. Ann Surg. 2016 Feb;263(2):234-9. doi: 10.1097/SLA.0000000000001504. PMID 26501704
- [Result] Usta TA, Gundogdu EC. The role of three-dimensional high-definition laparoscopic surgery for gynaecology. Curr Opin Obstet Gynecol. 2015 Aug;27(4):297-301. doi: 10.1097/GCO.0000000000000189. PMID 26107783
- [Result] Ozsoy M, Kallidonis P, Kyriazis I, Panagopoulos V, Vasilas M, Sakellaropoulos GC, Liatsikos E. Novice surgeons: do they benefit from 3D laparoscopy? Lasers Med Sci. 2015 May;30(4):1325-33. doi: 10.1007/s10103-015-1739-0. Epub 2015 Mar 15. PMID 25772250
- [Result] Ashraf A, Collins D, Whelan M, O'Sullivan R, Balfe P. Three-dimensional (3D) simulation versus two-dimensional (2D) enhances surgical skills acquisition in standardised laparoscopic tasks: a before and after study. Int J Surg. 2015 Feb;14:12-6. doi: 10.1016/j.ijsu.2014.12.020. Epub 2015 Jan 2. PMID 25560749
- [Result] Ko JK, Li RH, Cheung VY. Two-dimensional versus three-dimensional laparoscopy: evaluation of physicians' performance and preference using a pelvic trainer. J Minim Invasive Gynecol. 2015 Mar-Apr;22(3):421-7. doi: 10.1016/j.jmig.2014.11.007. Epub 2014 Nov 21. PMID 25461685
- [Result] Smith R, Schwab K, Day A, Rockall T, Ballard K, Bailey M, Jourdan I. Effect of passive polarizing three-dimensional displays on surgical performance for experienced laparoscopic surgeons. Br J Surg. 2014 Oct;101(11):1453-9. doi: 10.1002/bjs.9601. Epub 2014 Aug 18. PMID 25131843
- [Result] Alaraimi B, El Bakbak W, Sarker S, Makkiyah S, Al-Marzouq A, Goriparthi R, Bouhelal A, Quan V, Patel B. A randomized prospective study comparing acquisition of laparoscopic skills in three-dimensional (3D) vs. two-dimensional (2D) laparoscopy. World J Surg. 2014 Nov;38(11):2746-52. doi: 10.1007/s00268-014-2674-0. PMID 25002241
- [Result] Marcus HJ, Hughes-Hallett A, Cundy TP, Di Marco A, Pratt P, Nandi D, Darzi A, Yang GZ. Comparative effectiveness of 3-dimensional vs 2-dimensional and high-definition vs standard-definition neuroendoscopy: a preclinical randomized crossover study. Neurosurgery. 2014 Apr;74(4):375-80; discussion 380-1. doi: 10.1227/NEU.0000000000000249. PMID 24220007